CLINICAL TRIAL: NCT06156592
Title: Prospective Observational Study to Compare Hemodynamic Alterations in Severe Aortic Stenosis and Severe Mitral Regurgitation After High Spinal Anesthesia in Patients Undergoing Aortic Valve and Mitral Valve Replacement Surgery
Brief Title: Post Spinal Hemodynamic Changes in Aortic Stenosis and Mitral Regurgitation by VIS Index and Echocardiography
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: HS25925
Record Dates: First submitted 2023-09-24; First posted 2023-12-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-10

CONDITIONS: Severe Aortic Valve Stenosis; Severe Mitral Valve Regurgitation
Keywords: mitral valve replacement; aortic valve replacement; spinal anesthesia; echocardiographic monitoring; aortic stenosis; mitral regurgitation
MeSH Terms: conditions — Aortic Valve Stenosis; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe aortic stenosis group: Patients with severe aortic stenosis who are undergoing open aortic valve replacement under high spinal in combination with light general anesthesia.
  Interventions: Procedure: Cardiac valve replacement surgery under high spinal anesthesia combined with light general anesthesia
- Severe mitral regurgitation group: Patients with severe mitral regurgitation who are undergoing open mitral valve replacement under high spinal in combination with light general anesthesia.
  Interventions: Procedure: Cardiac valve replacement surgery under high spinal anesthesia combined with light general anesthesia

INTERVENTIONS:
Procedure: Cardiac valve replacement surgery under high spinal anesthesia combined with light general anesthesia — Before induction of general anesthesia, a high spinal anesthesia will be given using 37.5 mg of 0.75% heavy bupivacaine with 20 mcg fentanyl and 250 mcg epimorphine in sitting position at the lumbar intervertebral spaces between the L2-3 or L3-4 vertebrae. Patients will lie supine immediately afterwards, and sensory loss to ice will be performed every 15 seconds. Subsequently, the patient will be placed in 15-degree Trendelenburg (ensured by clinometer). Following general anesthesia will be induced and trachea will be intubated after 5 ml of 4% lignocaine spray on vocal cords and trachea. Hemodynamics will be aimed at MAP between 65-100 mmHg and heart rate between 50-100 beats /min by use of various inotropic, inodilators and vasoactive cardiac drugs based on anesthesiologists' clinical judgement.

SUMMARY:
This study will assess hemodynamic changes induced after spinal anesthesia by evaluating vasopressor inotropic requirements and variations in echocardiographic parameters in patients having severe aortic stenosis or severe mitral regurgitation undergoing aortic or mitral valve replacement surgery.

DETAILED DESCRIPTION:
Spinal anesthesia (SA) involves injecting local anesthetic into the intrathecal space. Since it was first described, understanding of the physiology and pharmacology of drugs acting within the subarachnoid space has improved. Physiological changes observed following SA are believed to be attributed to their blockade of peripheral and cardiac sympathetic fibers. The changes in cardiac output (CO) observed following SA were originally thought to be explained by the 'pre-load reduction' theory that describes a decrease in CO resulting from reduced venous return leading to arterial hypotension. However, this theory was questioned due to failed attempts to avoid SA induced hypotension by three preventative techniques: preloading with crystalloids or colloids, lower limb compression, and lateral tilt maneuvers (1). Additional studies and subsequent data led to further questioning of the pre-load reduction theory and supported a shift to an 'after-load reduction' theory. This proposes that hypotension following SA is a result of sympathetic blockade causing arterial dilatation (1,2). With this knowledge, it has traditionally been taught to avoid SA in severe aortic stenosis (AS) for risk of decreased coronary perfusion, while SA has been considered safe, or even beneficial in those with severe mitral regurgitation (MR). However, there is a paucity of real time evidence to help support these claims. Furthermore, individuals with experience in performing SA in patients with severe AS and/or MR have questioned the hemodynamic effects that are traditionally described (3).

With advancements in echocardiographic techniques, point of care ultrasound has emerged in critical care to become the standard for evaluating hemodynamic changes observed in hemodynamic instability or cardiovascular collapse (4). This provides an opportunity to assess CO, and its associated parameters including venous return, preload, afterload, and contractility, in real time. With this tool, one can compare the hemodynamic changes in patients with AS or MR before and after high SA given for their cardiac surgery for valve replacements or repair (AVR or MVR).

Hypothesis and Study Objectives:

This study may provide real time information to support or challenge traditional understanding of the hemodynamic changes seen following SA in those with severe AS or severe MR. Since, hemodynamic stability is goal in all patients after any type of anesthesia, the primary objective is to compare requirement of vasopressors, inotropes, and inodilators required to maintain desired hemodynamic goals (Mean arterial pressure 65-100 mmHg and HR 50-100/min) and to observe and compare hemodynamics alteration by using echocardiographic parameters of venous return, cardiac index (CI), preload, afterload, and cardiac contractility using myocardial performance index (Tei index) (5) before and after high SA in patients having predominant severe AS or MR. Furthermore, subgroup analysis will be conducted to compare hemodynamic parameters and medication requirements to meet target hemodynamic goals among patients with preserved and reduced left ventricular systolic function (for AS reduced LVEF < 50 %, for MR reduced LVEF < 60%).

Methodology:

This prospective observational study will be conducted at St. Boniface Hospital, Winnipeg, Canada. All adult patients above 18 years of age, irrespective of their gender, ASA physical status, and LVEF requiring SA up to T1-2 level block with light general anesthesia (GA) for their surgical procedures of AVR or MVR will be included. Exclusion criteria: Mixed valvular lesion (more than mild AR or MS), redo cardiac surgery, not eligible for fast tracking (i.e., anticipated post-surgical extubation time more than 10 hours (6) of successful uncomplicated surgery, unable of laying supine in 15-degree Trendelenburg, hypoxic patients (SaO2 less than 94% on room air), difficult airway requiring awake intubation, patients receiving dialysis, contraindication for transesophageal echo (TEE) or spinal anesthesia, significant deformity of thoracic and lumbar spine and poor TTE windows for data acquisition. Patients undergoing associated CABG for single vessel and without significant regional wall motion abnormalities on echo (no more than 3 segment involvement), will be included. Patients will be consented for the study once eligible participants are identified in the cardiac anesthesia PAC clinic.

All TTE parameters will be recorded in the apical 4 and 5 chamber views with a Phillips echo Apiq 7 machine. The following baseline echo parameters to be recorded will be linear dimensions of tricuspid valve (TV) and mitral valve (MV) annulus in 4C view left ventricular outflow tract (LVOT) in Plax view, and LVEF in apical 4C view and LV short axis view. The linear dimensions of TV and MV annulus and LVOT will also be confirmed on TEE views and final measurement will be relied on more crisp views. At baseline echo and repeat assessments, the parameters to be recorded will be velocity time integral (VTI) of LVOT, MV, TV, tricuspid annular plane systolic excursion (TAPSE) and mitral annular plane systolic excursion (MAPSE) on M-Mode, and tissue doppler imaging (TDI) of lateral TV and MV annulus. To calculate LV Tei index Doppler time intervals measured from MV inflow and LVOT Doppler tracings, as described by Tei and co-workers will be used (5). Tei index will also be calculated from TDI interrogation using 1.5 mm sample volume from lateral MV and TV for LV and RV (6,7). For LV Tei index mean of values from TDI and PWD will be used for analysis. No correction for HR variability will be applied for Tei index below HR 100/min (8). In patients with atrial fibrillation (AF), "pre ejection period (PEP)-derived MPI (Tei index)" will be calculated since the loss of mechanical atrial function does not allow measurement of isovolumic contraction time (IVCT) (9). On TEE, a mid-esophageal (ME) 4 and Deep TG views will be used post intubation for same Doppler and M mode parameters.

Among cardiac medications only beta blockers will be continued on am of surgery. Once in the operating room, all patients will have two intravenous lines, ECG, arterial line, central venous line, pulse oximetry, defibrillator pads, cerebral oximetry and patient state index (PSi) by Masio monitored. During the study period, Ringer's Lactate will be infused at a rate of 600ml/hr (100 ml infusion drive line and 500 ml/hr second iv line which will also be used for drug boluses). Intraoperative hemodynamic parameters will be automatically recorded by computer interphase system with Philips monitors. A high spinal will be given using 37.5 mg of 0.75% bupivacaine heavy with 20 mcg fentanyl and 250 mcg epimorphine in sitting position at the lumbar intervertebral spaces between the L2-3 or L3-4 vertebrae with 25 G Whitacre or Quincke needle. Patients will lie supine immediately afterwards, and sensory loss to ice will be performed every 15 seconds. Echo parameters with TTE will be recorded before spinal, at sensory loss between T10-12 in flat supine. Subsequently, the patient will be placed in 15-degree Trendelenburg (ensured by clinometer) and once sensory loss between T4-T8 occurs, a third TTE recording will be performed while patient being preoxygenated in preparation for GA. Afterwards, patients will be induced by general anesthesia (GA) in the Trendelenburg position, and a fourth echo recording will be performed by TEE under GA after putting CVL and first CVP reading is taken by keeping transducer at heart level in the mid axillary line. Final fifth TEE echo parameters will be recorded in final surgical position which will be flat supine with back up to 5 degrees.

A change in SBP or MAP equal to or less than 10% mmHg and HR equal to or less than 10% beats/min from readings before incision within one minute of skin incision and sternotomy will be considered "no response" and an effective sensory block unto T1.

General anesthesia will be induced by 0.02-0.03 mg/Kg midazolam (maximum 2 mg), 0.2-0.4 mg/Kg ketamine (maximum 20 mg), 0.3-0.5 mcg/Kg sufentanil, titrated dose of 1-3 mg/Kg propofol to loss of eye reflex, and rocuronium 1.0-1.2 mg/kg. Intubation will be preceded with 5 ml of 4% lignocaine spray on the vocal cords and in trachea. Post intubation anesthesia will be maintained by 50% oxygen with sevoflurane 1-2 % end tidal value titrated to PSI 30-50 on Massimo monitor, volume control ventilation targeting EtCO2 goal of 35-40 mmHg. During the study period target hemodynamics will be aimed at MAP between 65-100 mmHg and heart rate between 50-100 beats /min by use of various inotropic, inodilators and vasoactive cardiac drugs based on anesthesiologists' clinical judgement. Total dose of boluses and infusions of these drugs used during study period will be recorded for comparison as cumulated modified vasopressor inotropic inodilator score index during pre CPB, on CPB and post CPB period till patient leaves the operation room. This will be calculated as follows:

Total modified VIS score (pre CPB or on CPB or post CPB) = (total dopamine in mcg ) + (total dobutamine in mcg) + (10 x total milrinone in mcg) + (10,000 x total vasopressin unit) + (100 x total norepinephrine in mcg) + ( 100 x total epinephrine dose mcg) + (100 x total ephedrine dose in mg) + (10 x total phenylephrine dose in mcg) VIS index = Total modified VIS score / (weight in Kg x time in minutes)

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age, irrespective of their gender or ASA physical status
* With severe aortic stenosis or mitral regurgitation
* Undergoing elective aortic or mitral valve repair or replacement
* Eligible for spinal anesthesia up to T1-2 level block for their surgical procedure.
* Able to provide written informed consent

Exclusion Criteria:

* Contraindications to the administration of spinal anesthesia such as pre-existing coagulopathy, local sepsis at the site of insertion
* Hypoxic (SaO2 < 95%) on room air
* Unable to lie flat and with 15-degree trendelenburg
* The apical four and five chamber window is not accessible on trans-thoracic echocardiography
* Difficult airway requiring awake intubation
* On dialysis
* Redo-valve surgery
* Mixed valvular lesions (more than mild AR or MS)
* Requiring more than one CABG or CPB duration more than 180 minutes
* More than 3 segment Regional Wall Motion Abnormalities
* Severe spine disorders

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to St. Boniface Hospital, Winnipeg, Canada, a tertiary care hospital, for elective aortic or mitral valve repair over the period Oct 2023 to December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-26 (Actual); Study Completion 2025-10-26 (Actual)

PRIMARY OUTCOMES:
To compare total inotropic, inodilators and vasopressor drug requirements by calculating the vasoactive-inotropic score (VIS) Index to maintain target stable hemodynamics in both groups | From spinal drug injection to the starting of cardiopulmonary bypass (CPB), during CPB surgery and post CPB up to the time when patient leaves operation room
  Total modified VIS score (pre CPB or on CPB or post CPB) = (total dopamine in mcg ) + (total dobutamine in mcg) + (10 x total milrinone in mcg) + (10,000 x total vasopressin unit) + (100 x total norepinephrine in mcg) + ( 100 x total epinephrine dose mcg) + (100 x total ephedrine dose in mg) VIS index = Total modified VIS score / (weight in Kg x time in minutes)
To compare changes in right and left ventricular myocardial performance index (Tei) in both groups | Baseline pre-spinal, 2 minutes post spinal flat supine, 5 min post spinal trendelenburg 15 degree,10 minutes post general anesthesia at opening CVP pressure in trendelenburg 15 degree, 2 minute post surgical position flat supine with 5 degree back up
  Tei index for the left ventricle will be derived using Doppler interrogation MV and left ventricular outflow tract (LVOT) blood flows and for both RV and LV by tissue Doppler interrogation of TV and MV lateral annular plane motion on echocardiography in both groups
To compare changes in Left Ventricular Outflow Tract (LVOT) Cardiac Index (CI) in both groups | Baseline pre-spinal, 2 minutes post spinal flat supine, 5 min post spinal trendelenburg 15 degree,10 minutes post general anesthesia at opening CVP pressure in trendelenburg 15 degree, 2 minute post surgical position flat supine with 5 degree back up
  LVOT cardiac index will be derived pulse wave Doppler interrogation of LVOT flow, 2 dimensional LVOT area and heart rate by echocardiography

SECONDARY OUTCOMES:
Subgroup analysis of patients with preserved Left Ventricular Ejection Fraction (LVEF) and reduced LVEF for comparison of Tei index of right ventricle, and left ventricle, TAPSE, MAPSE and LVOT CI by echocardiography and VIS index to maintain target he | Similar pre-defined time points for echocardiography readings and VIS index durations as for primary end points.
  Subgroup division will be done among all patients irrespective of primary valvular lesion based on LVEF which will be considered reduced if less than 50% in aortic stenosis and less than 60% in mitral regurgitation
Assessment and determination of changes in other echocardiographic hemodynamic parameters of preload, after load after high spinal anesthesia in severe AS and severe MR and their comparison to baseline and between these two valvular pathologies. | Baseline pre-spinal, 2 minutes post spinal flat supine, 5 min post spinal trendelenburg 15 degree,10 minutes post general anesthesia at opening CVP pressure in trendelenburg 15 degree, 2 minute post surgical position flat supine with 5 degree back up
  Echocardiographic measurements of TV flow, MV flow, and calculated preload and afterload from LV dimensions and CVP and arterial pressures will be derived using Laplace equation
Assessment and determination of changes in other echocardiographic parameters of RV contractility after high spinal anesthesia in severe AS and severe MR and their comparison to baseline and between these two valvular pathologies. | Baseline pre-spinal, 2 minutes post spinal flat supine, 5 min post spinal trendelenburg 15 degree,10 minutes post general anesthesia at opening CVP pressure in trendelenburg 15 degree, 2 minute post surgical position flat supine with 5 degree back up
  Echocardiographic measurements of TV annular plane systolic excursion (TAPSE) by M-mode application
Assessment and determination of changes in other echocardiographic parameters of LV contractility after high spinal anesthesia in severe AS and severe MR and their comparison to baseline and between these two valvular pathologies. | Baseline pre-spinal, 2 minutes post spinal flat supine, 5 min post spinal trendelenburg 15 degree,10 minutes post general anesthesia at opening CVP pressure in trendelenburg 15 degree, 2 minute post surgical position flat supine with 5 degree back up
  Echocardiographic measurements of MV annular plane systolic excursion (MAPSE) by M-mode application
Comparison of pulse oximetry and cerebral oximetry changes during study period between AS and MR patients | Baseline, at echo reading time points, and every 15 minutes afterwards to the end of surgery in both the groups
  This will be done using pulse oximeter and cerebral oximeter by Masimo monitor
Comparison of any complications in both group and subgroups during study period | From spinal drug injection to the starting of cardiopulmonary bypass (CPB), during CPB surgery and post CPB up to the time 48 hours in cardiac intensive care unit
  Any arrhythmia, hemodynamic episode outside target, spinal anesthesia complications, any unforeseen complication

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Arya, MD, FRCPC, Principal Investigator — SBGH, University of Manitoba, Winnipeg, Canada
Locations (1):
- Department of Anesthesiology, Perioperative and Pain Medicine, SBGH, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson E. 'Advances in understanding and management in obstetric anaesthesia': The great myth of our times. Indian J Anaesth. 2017 Apr;61(4):285-288. doi: 10.4103/ija.IJA_209_17. No abstract available. PMID 28515514
- [Background] Langesaeter E, Rosseland LA, Stubhaug A. Continuous invasive blood pressure and cardiac output monitoring during cesarean delivery: a randomized, double-blind comparison of low-dose versus high-dose spinal anesthesia with intravenous phenylephrine or placebo infusion. Anesthesiology. 2008 Nov;109(5):856-63. doi: 10.1097/ALN.0b013e31818a401f. PMID 18946298
- [Background] Bhat I, Arya VK, Mandal B, Jayant A, Dutta V, Rana SS. Postoperative hemodynamics after high spinal block with or without intrathecal morphine in cardiac surgical patients: a randomized-controlled trial. Can J Anaesth. 2021 Jun;68(6):825-834. doi: 10.1007/s12630-021-01937-z. Epub 2021 Feb 9. PMID 33564993
- [Background] Arya VK, Al-Moustadi W, Dutta V. Cardiac output monitoring - invasive and noninvasive. Curr Opin Crit Care. 2022 Jun 1;28(3):340-347. doi: 10.1097/MCC.0000000000000937. Epub 2022 Mar 11. PMID 35275876
- [Background] Tei C, Ling LH, Hodge DO, Bailey KR, Oh JK, Rodeheffer RJ, Tajik AJ, Seward JB. New index of combined systolic and diastolic myocardial performance: a simple and reproducible measure of cardiac function--a study in normals and dilated cardiomyopathy. J Cardiol. 1995 Dec;26(6):357-66. PMID 8558414
- [Background] Cheng DC. Fast track cardiac surgery pathways: early extubation, process of care, and cost containment. Anesthesiology. 1998 Jun;88(6):1429-33. doi: 10.1097/00000542-199806000-00002. No abstract available. PMID 9637632
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Poulsen SH, Nielsen JC, Andersen HR. The influence of heart rate on the Doppler-derived myocardial performance index. J Am Soc Echocardiogr. 2000 May;13(5):379-84. doi: 10.1016/s0894-7317(00)70007-1. PMID 10804435
- [Background] Su HM, Lin TH, Hsu PC, Chu CY, Lee WH, Lee CS, Lai WT, Sheu SH, Voon WC. Myocardial performance index derived from preejection period: a novel and feasible parameter in evaluation of cardiac performance in patients with permanent atrial fibrillation. Echocardiography. 2011 Nov;28(10):1081-7. doi: 10.1111/j.1540-8175.2011.01491.x. Epub 2011 Aug 19. PMID 22077881